CLINICAL TRIAL: NCT02774876
Title: An Open-label, Randomized, Four-way, Cross-over Study to Examine the Efficacy of Single-hormone Closed-loop System in Regulating Glucose Levels in Adults With Type 1 Diabetes Following Meals of Various Macronutrient Contents: a Pilot Study
Brief Title: Closed-loop Control of Postprandial Glucose Levels After Meals With Different Macronutrients Content in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-Macro
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop system; Artificial pancreas; Glucose control; Meal
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Carbohydrate meal (Active Comparator)
  Interventions: Device: Patient's insulin pump; Drug: Insulin; Device: Dexcom G4 Platinum glucose sensor; Other: Single-hormone closed-loop
- Carbohydrate + fat meal (Active Comparator)
  Interventions: Device: Patient's insulin pump; Drug: Insulin; Device: Dexcom G4 Platinum glucose sensor; Other: Single-hormone closed-loop
- Carbohydrate + protein meal (Active Comparator)
  Interventions: Device: Patient's insulin pump; Drug: Insulin; Device: Dexcom G4 Platinum glucose sensor; Other: Single-hormone closed-loop
- Carbohydrate + fat + protein meal (Active Comparator)
  Interventions: Device: Patient's insulin pump; Drug: Insulin; Device: Dexcom G4 Platinum glucose sensor; Other: Single-hormone closed-loop

INTERVENTIONS:
Device: Patient's insulin pump — The patient's insulin pump will be used to regulate glucose levels.
Drug: Insulin — Patient's usual fast-acting insulin analog will be used.
Device: Dexcom G4 Platinum glucose sensor — The Dexcom G4 Platinum glucose sensor will be used to measure glucose levels.
Other: Single-hormone closed-loop — Interventions will be undertaken 1 to 5 days after sensor insertion. Subjects will be admitted at IRCM at 6:30 am in a fasting state. At 7:00, single-hormone closed-loop will be initiated. At 8:00, if glucose levels are between 3.5 and 12.5 mmol/L, the meal will be served. Patients will have 20 minutes to consume the meal. If glucose levels are not in this target range, the meal will be delayed for a maximum of 45 minutes. If after 45 minutes, glucoses levels are still not between 3.5 and 12.5 mmol/L, the test will be cancelled and rescheduled. The test meals will be: 1) 75g of CHO; 2) 75g of CHO + 35g of protein; 3) 75g of CHO + 35g of fat; or 4) 75g of CHO + 35g of protein + 35g of fat. The intervention day will end at 13:00.

SUMMARY:
Carbohydrates are the main determinant of post-meal glucose excursion. However, fat and protein have been shown to also impact the postprandial glucose control, adding to the complexity of meal insulin calculation. Few studies have looked at the effect of macronutrients other than carbohydrates on postprandial glucose excursions with the closed-loop strategy. The objective of this study is to test whether the single-hormone closed-loop strategy can achieve similar post-meal glucose control with meals with a fixed carbohydrate content, but high in protein and/or fat when compared to a meal with a fixed carbohydrate content only.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months and currently using fast-acting insulin analog (Lispro, Aspart or Guilisine).
4. Last (less than 3 months) HbA1c ≤ 10%.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Ongoing pregnancy.
4. Severe hypoglycemic episode within 1 month of screening.
5. Agents affecting gastric emptying (Motilium®, Prandase®, all GLP-1 analogs) as well as oral anti-diabetic agents (Metformin, SGLT-2 inhibitors and DPP-4 inhibitors) if not at a stable dose for 3 months. Otherwise, these medications are acceptable and will be kept stable during the entire protocol.
6. Oral steroids unless patients present a low stable dose (e.g. 10 mg or less of prednisone per day or physiological doses, less than 35 mg/day, of hydrocortisone Cortef®). Inhaled steroids at stable dose in the last month are acceptable.
7. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator (e.g. unstable psychiatric condition).
8. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, follow algorithm's suggestions, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve of sensor glucose levels | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.

SECONDARY OUTCOMES:
Mean sensor glucose levels | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Peak glucose excursion | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Time to peak glucose | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Percentage of time of sensor glucose concentrations between 3.9 and 7.8 mmol/L | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Percentage of time of sensor glucose concentrations between 3.9 and 10 mmol/L | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Percentage of time of sensor glucose concentrations above 10 mmol/L | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Percentage of time of sensor glucose concentrations above 13.9 mmol/L | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Total insulin delivery | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Standard deviation of glucose levels | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.
Coefficient of variation of glucose levels | The outcome measure will be calculated over the 5 hours following the breakfast meal given on the single-hormone closed-loop intervention. The 5-hour period is from 8:00 to 13:00.

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No